CLINICAL TRIAL: NCT04116567
Title: Lung Ultrasonography for the Assessment of Perioperative Atelectasis After Laparoscopic Gynecologic Oncologic Surgery
Brief Title: Lung Ultrasonography After Laparoscopic Gynecologic Surgery
Acronym: LUS-LPS
Status: Completed | Type: Observational
Sponsor: SONNINO CHIARA (Other)
Responsible Party: Sponsor-Investigator, SONNINO CHIARA, Registered Anesthesiologist, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Organization: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Other Study IDs: 2560
Record Dates: First submitted 2019-07-27; First posted 2019-10-04 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Pulmonary Atelectasis
Keywords: Pulmonary Atelectasis; Lung Ultrasound; Laparoscopic Surgery
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study evaluates the influence of surgical and anesthesia-related variable on atelectasis formation during laparoscopic gynecologic oncologic surgery by lung ultrasound.

DETAILED DESCRIPTION:
Approximately 50% of patients undergoing general anesthesia are hypoxemic. Anaesthesia, paralysis, high concentrations of oxygen, inadequate level of PEEP, capnoperitoneum, Trendelenburg position all result in persistent atelectasis. Lung ultrasound is a safe and accurate bedside tool useful to study lung aeration. The aim of the investigator's study was to assess the impact of general anesthesia and laparoscopic gynecologic oncologic surgery on post-operative atelectasis and related oxygenation changes using lung ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 yo undergoing laparoscopic surgery for gynecologic surgery who provide written informed consent.

Exclusion Criteria:

* age < 18 yo;
* pregnancy;
* refused to partecipate;
* known pulmonary metastasis;
* preexisting pulmonary conditions (COPD, pleural effusion, pulmonary consolidations, lung edema, pulmonary embolism);
* anesthesia with mechanical ventilation in the 2 weeks.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients >18yo undergoing laparoscopy for ginecologic oncologic surgery willing to participate to the study
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2018-10-03 (Actual); Primary Completion 2018-10-03 (Actual); Study Completion 2019-06-28 (Actual)

PRIMARY OUTCOMES:
Assess if LUS score measured after surgery is higher that LUS score measured before induction of anesthesia | The outcome will be measured 10 minutes after extubation
  Each lung will be divided in 6 areas and a score from 0 to 3 will be assigned to each field depending on the loss of aereation detected by ultrasound. LUS score will range between 0 and 36. Lung ultrasound will be performed before induction of anesthesia and 10 minutes after extubation.
Correlation between the increase of LUS score after surgery and surgical or anesthesia-related variables. | The outcome will be measured 10 minutes after extubation
  Logistic regression will be applied to consider the correlation between Delta LUS and the following variables:
  * lenght of surgery
  * duration of pneumoperitoneum
  * angle of Trendelenburg potision
  * duration of mechanical ventilation
  * intraoperative fluids
  * duration of apnea from induction to intubation

CONTACTS AND LOCATIONS:
Overall Officials: Luciano Frassanito, MD, Principal Investigator — IRCCS Fondazione Universitaria Policlinico Agostino Gemelli; Gaetano Draisci, MD, PhD, Study Director — IRCCS Fondazione Universitaria Policlinico Agostino Gemelli
Locations (1):
- IRCCS Fondazione Policlinico Universitario Agostino Gemelli, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided